CLINICAL TRIAL: NCT04080570
Title: Remote Physician Care for Home Hospital Patients: A Randomized Controlled Trial
Brief Title: Remote Physician Care for Home Hospital Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Levine, Instructor in Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P002583
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Infection; Heart Failure; Chronic Obstructive Pulmonary Disease; Asthma; Gout Flare; Chronic Kidney Diseases; Hypertensive Urgency; Atrial Fibrillation Rapid; Anticoagulants; Increased
Keywords: home hospital; hospital at home; hospital in the home
MeSH Terms: conditions — Infections; Heart Failure; Pulmonary Disease, Chronic Obstructive; Asthma; Renal Insufficiency, Chronic; Hypertensive Crisis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Visit (Experimental): After an initial physical in-home visit, the physician will see home hospitalized patients by facilitated video each day.
  Interventions: Other: Remote Visit
- In-Home Visit (No Intervention): The physician will see home hospitalized patients physically in their homes each day, as is usual care.

INTERVENTIONS:
Other: Remote Visit — After an initial in-home visit, the physician will see home hospitalized patients by facilitated video.
  Arms: Remote Visit

SUMMARY:
This study examines the implications of providing remote physician care to home hospitalized patients compared to usual home hospital care with in-person/in-home physician visits.

DETAILED DESCRIPTION:
Home hospital care is hospital-level care at home for acutely ill patients. In multiple publications, home hospital care delivered cost-effective, high-quality, excellent experience care with similar quality and safety as traditional hospital care. Most home hospital models require a licensed independent practitioner to see their patients physically in their home.

To further improve the efficiency and scalability of home hospital care, the investigators propose to test remote care, where the physician would provide care via a video interaction, instead of in-home/in-person care. The investigators propose a non-inferiority evaluation of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Resides within either a 5-mile or 20 minute driving radius of emergency department
* Has capacity to consent to study OR can assent to study and has proxy who can consent
* >= 18 years-old
* Can identify a potential caregiver who agrees to stay with patient for first 24 hours of admission. Caregiver must be competent to call care team if a problem is evident to her/him. After 24 hours, this caregiver should be available for as-needed spot checks on the patient. This criterion may be waived for highly competent patients at the patient and clinician's discretion.
* Primary or possible diagnosis of cellulitis, heart failure, complicated urinary tract infection, pneumonia, COPD/asthma, other infection, chronic kidney disease, malignant pain, diabetes and its complications, gout flare, hypertensive urgency, previously diagnosed atrial fibrillation with rapid ventricular response, anticoagulation needs, or a patient who desires only medical management that requires inpatient admission, as determined by the emergency room team.

Exclusion Criteria:

* Undomiciled
* No working heat (October-April), no working air conditioning if forecast > 80°F (June-September), or no running water
* On methadone requiring daily pickup of medication
* In police custody
* Resides in facility that provides on-site medical care (e.g., skilled nursing facility)
* Domestic violence screen positive
* Acute delirium, as determined by the Confusion Assessment Method2
* Cannot establish peripheral access in emergency department (or access requires ultrasound guidance, unless point-of-care ultrasound is available)
* Secondary condition: end-stage renal disease on hemodialysis, acute myocardial infarction, acute cerebral vascular accident, acute hemorrhage
* Primary diagnosis requires multiple or routine administrations of intravenous narcotics for pain control
* Cannot independently ambulate to bedside commode, unless home-based aides are available
* As deemed by on-call MD, patient likely to require any of the following procedures: computed tomography, magnetic resonance imaging, endoscopic procedure, blood transfusion, cardiac stress test, or surgery
* High risk for clinical deterioration
* Home hospital census is full

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2019-08-03 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Adverse events, # | From date of admission to date of discharge (except for 30-day mortality), an expected average of 4 days
  The per patient count of adverse events, including fall, delirium, potentially preventable venous thromboembolism, new pressure ulcer, thrombophlebitis at peripheral IV site, catheter-associated urinary tract infection, new Clostridium difficile, new methicillin-resistant Staphylococcus aureus, new arrhythmia, hypokalemia, acute kidney injury, transfer back to hospital, mortality (unplanned) during admission, mortality (unplanned) 30-day post-discharge.

SECONDARY OUTCOMES:
Unplanned readmission after index admission, y/n | Day of discharge to 30 days later
Picker experience questionnaire, score | Day of discharge, an expected average of 4 days
  Score between 0 and 15, with higher scores signifying better experience
Global experience, score | Day of discharge, an expected average of 4 days
  Score between 0 and 10, with higher scores signifying better experience

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Faulkner Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leff B, Burton L, Mader SL, Naughton B, Burl J, Inouye SK, Greenough WB 3rd, Guido S, Langston C, Frick KD, Steinwachs D, Burton JR. Hospital at home: feasibility and outcomes of a program to provide hospital-level care at home for acutely ill older patients. Ann Intern Med. 2005 Dec 6;143(11):798-808. doi: 10.7326/0003-4819-143-11-200512060-00008. PMID 16330791
- [Background] Cryer L, Shannon SB, Van Amsterdam M, Leff B. Costs for 'hospital at home' patients were 19 percent lower, with equal or better outcomes compared to similar inpatients. Health Aff (Millwood). 2012 Jun;31(6):1237-43. doi: 10.1377/hlthaff.2011.1132. PMID 22665835
- [Background] Montalto M. The 500-bed hospital that isn't there: the Victorian Department of Health review of the Hospital in the Home program. Med J Aust. 2010 Nov 15;193(10):598-601. doi: 10.5694/j.1326-5377.2010.tb04070.x. PMID 21077817
- [Background] Levine DM, Ouchi K, Blanchfield B, Diamond K, Licurse A, Pu CT, Schnipper JL. Hospital-Level Care at Home for Acutely Ill Adults: a Pilot Randomized Controlled Trial. J Gen Intern Med. 2018 May;33(5):729-736. doi: 10.1007/s11606-018-4307-z. Epub 2018 Feb 6. PMID 29411238
- [Background] Federman AD, Soones T, DeCherrie LV, Leff B, Siu AL. Association of a Bundled Hospital-at-Home and 30-Day Postacute Transitional Care Program With Clinical Outcomes and Patient Experiences. JAMA Intern Med. 2018 Aug 1;178(8):1033-1040. doi: 10.1001/jamainternmed.2018.2562. PMID 29946693
- [Derived] Levine DM, Paz M, Burke K, Beaumont R, Boxer RB, Morris CA, Britton KA, Orav EJ, Schnipper JL. Remote vs In-home Physician Visits for Hospital-Level Care at Home: A Randomized Clinical Trial. JAMA Netw Open. 2022 Aug 1;5(8):e2229067. doi: 10.1001/jamanetworkopen.2022.29067. PMID 36040741